CLINICAL TRIAL: NCT01899274
Title: Assessment of an Electronic Self-Management Tool on Glycemic Control in Teens With Type 1 Diabetes
Brief Title: Assessment of an iPhone Application on Glycemic Control in Type 1 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Collaborators: Thrasher Research Fund (Other); University Health Network, Toronto (Other); York University (Other)
Responsible Party: Principal Investigator, Mark Palmert, Head of Division of Endocrinology, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1000036524; 11054 (Other Grant/Funding Number: Thrasher Research Fund)
Record Dates: First submitted 2013-07-10; First posted 2013-07-15 (Estimated); Last update posted 2016-04-19 (Estimated); Status verified 2016-04

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- bant Group (Experimental): Subjects in the bant Group will receive care as usual, as well as an iPhone loaded with the bant iPhone application and a bluetooth enabled glucometer. Participants will have their A1C levels measured every 3 months (for 1 year), and also complete questionnaires/interviews relating to their diabetes management and lifestyle.
  Interventions: Device: bant iPhone application
- Control Group (No Intervention): Subjects in the control group will continue care as usual with their diabetes team, without supplementation of the bant application. Participants will have their A1C levels measured every 3 months (for 1 year), as well as complete questionnaires/interviews relating to their diabetes management and lifestyle.

INTERVENTIONS:
Device: bant iPhone application
  Arms: bant Group

SUMMARY:
The purpose of the study is to assess whether an electronic self-management tool, specifically an iPhone application entitled bant, can improve glycemic control in Adolescents who have Type 1 Diabetes Mellitus (T1DM).

DETAILED DESCRIPTION:
Type 1 Diabetes Mellitus (T1DM) is among the most common chronic diseases affecting children, adolescents and adults. While intensive patient self-management can optimize Blood Glucose (BG) to near-normal levels, it is a challenge for many TIDM patients to continuously achieve this. These difficulties are compounded in the adolescent population, who struggle with daily self-management and therefore may increase their risk of T1DM complications.

Due to this observation an electronic self-management tool, in the form of an iPhone application called bant, was developed. This app guides the analysis of BG data and suggests changes in treatment, while also using social network and rewards to encourage and reinforce self-care behaviors, such as frequent self-monitoring of blood glucose levels (SMBG). By primarily measuring changes in HbA1C levels, the study will assess if bant and its features are associated with improved glycemic control in the adolescents who use it.

ELIGIBILITY:
Inclusion Criteria:

* T1DM as defined by 2008 Canadian Diabetes Association (CDA,2008)guidelines, with duration ≥ 1 year
* Age 11-16 years, inclusive at enrollment in the trial
* 2 of the participant's last 3 A1C results prior to enrollment, including the most recent, falling between 8.0% - 10.5%
* Have been followed for at least 6 months in the current diabetes clinic

Exclusion Criteria:

* Non-English speaking adolescents as the version of bant being used in the randomized control trial (RCT) is only offered in English at this time.

Ages: 11 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 92 (Actual)
Dates: Start 2013-07; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Changes in Hemoglobin A1C levels | 12 month RCT duration
  Hemoglobin A1C levels are a common and important measure of diabetes control, and will be collected at baseline, regular 3-month research follow-ups, a final 12-month research visit. Primary Outcome will be based on comparison of A1C values at baseline to A1C values at RCT completion (12 months).
  In order to assess the potential durability of the intervention, A1C values will also be recorded (from clinical visits) 6-months and 12-months post-RCT completion.

SECONDARY OUTCOMES:
Hypoglycemic Events | 12 month RCT duration
  Hypoglycemic events will be measured at baseline, and every following 3 months (for 1 year). These will include both severe hypoglycemic events (requiring assistance of another individual with a BG <2.8 mmol/l and/or reversal of symptoms with oral or intravenous carbohydrate/glucose) and mild hypoglycemic events (BG <3.4mmol/L).
Self-Efficacy | 12 month RCT duration
  Participant Self-Efficacy will be measured using verified survey and questionnaire tools. Data will be collected at baseline and every following 3 months (for 1 year).
Self-Care Behaviour | 12 month RCT duration
  Self-Care Behaviour will be measured using verified survey and questionnaire tools. Data will be collected at baseline and every following 3 months (for 1 year).
Treatment Adherence | 12 month RCT duration
  Participant Treatment Adherence will be measured using verified survey and questionnaire tools. Data will be collected at baseline and every following 3 months (for 1 year).
Quality of Life | 12 month RCT duration
  Participant Quality of Life will be measured using verified survey and questionnaire tools. Data will be collected at baseline and every following 3 months (for 1 year).
bant Component Usage | 12 month RCT duration
  Usage rates of various bant components, such as social networking and rewards, will be monitored and correlated with changes in primary and secondary outcome measures.

CONTACTS AND LOCATIONS:
Overall Officials: Mark R Palmert, M.D., Ph.D., Principal Investigator — The Hospital for Sick Children
Locations (2):
- Canada (2):
  - Trillium Health Partners, Mississauga, Ontario
  - The Hostpital for Sick Children, Toronto, Ontario

REFERENCES:
- [Result] Cafazzo JA, Casselman M, Hamming N, Katzman DK, Palmert MR. Design of an mHealth app for the self-management of adolescent type 1 diabetes: a pilot study. J Med Internet Res. 2012 May 8;14(3):e70. doi: 10.2196/jmir.2058. PMID 22564332
- [Derived] Goyal S, Nunn CA, Rotondi M, Couperthwaite AB, Reiser S, Simone A, Katzman DK, Cafazzo JA, Palmert MR. A Mobile App for the Self-Management of Type 1 Diabetes Among Adolescents: A Randomized Controlled Trial. JMIR Mhealth Uhealth. 2017 Jun 19;5(6):e82. doi: 10.2196/mhealth.7336. PMID 28630037